CLINICAL TRIAL: NCT07184320
Title: The Impact of AI-Based Video Education on Denture Care and Oral Health-Related Quality of Life Among Older Adults: A Nursing-Prosthodontic Collaborative Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sherif Aly Sadek (Other)
Collaborators: Gulf Medical University (Other)
Responsible Party: Sponsor-Investigator, Sherif Aly Sadek, Associate Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-COD-FAC-06-Aug-2025
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Complete Edentulism; Partial Denture; Partial Edentulism in the Maxilla or in the Mandible
Keywords: Digital Health Education; Denture Care; Patient Education; Interdisciplinary Care; Prosthodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-Based Video Education (Experimental): Participants will receive structured AI-based video education on denture care
  Interventions: Behavioral: AI-Based Video Education on Denture Care
- Conventional Oral Health Instruction (Active Comparator): Participants will receive conventional chairside verbal oral health instruction from the prosthodontic team on denture care
  Interventions: Behavioral: Conventional Oral Health Instruction

INTERVENTIONS:
Behavioral: AI-Based Video Education on Denture Care — The intervention consists of an AI-based educational video module, approximately 8 minutes in duration, designed to improve denture care practices. It uses step-by-step, visually engaging demonstrations with AI-guided narration to enhance understanding, recall, and adherence.
  Arms: AI-Based Video Education
Behavioral: Conventional Oral Health Instruction — Participants in the control group will receive conventional oral health education delivered verbally and chairside by the prosthodontic team. The standardized instruction includes information on denture hygiene techniques, appropriate storage of dentures overnight, mucosal care
  Arms: Conventional Oral Health Instruction

SUMMARY:
To assess the effectiveness of AI-based educational videos in improving patient-reported oral health outcomes.

DETAILED DESCRIPTION:
This study adopts a two-arm, parallel-group randomised controlled trial (RCT) design to compare the effectiveness of AI-based video education versus conventional oral health instruction in improving denture care knowledge, patient satisfaction, and oral health-related quality of life among older adults wearing removable prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 50 years old.
* Patients are removable denture users.
* Patients can consent.
* Patients who completed follow-up.

Exclusion Criteria:

* Patients with cognitive impairment.
* Participants are currently rehabilitated with fixed prostheses.
* Patients received prior structured education in the last 6 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Oral Health-Related Quality of Life (OHIP-14 Score) | Baseline, immediately post-intervention, 1 month, 2 months, and 3 months
  The primary outcome is the mean change in OHIP-14 total score from baseline to follow-up assessments.

SECONDARY OUTCOMES:
Change in Denture Care Knowledge Retention Score | Baseline, immediately post-intervention, 1 month, 2 months, and 3 months
  Measured using a structured denture care knowledge quiz assessing correct cleaning frequency, storage methods, avoidance of harmful practices, recognition of poor fit, and oral hygiene procedures.
Patient Satisfaction with Educational Method | Immediately post-intervention, 1 month, 2 months, and 3 months
  Measured using a 5-point Likert scale questionnaire evaluating clarity, usefulness, acceptability, and confidence in applying denture care practices after receiving the assigned intervention (AI-based video or conventional oral instruction).
Compliance with Denture Hygiene Practices | 1 month, 2 months, and 3 months post-intervention
  Assessed with a structured self-reported checklist of daily denture care practices, including cleaning frequency, storage behaviour, and oral mucosal care.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulf Medical University, Ajman, Ajman Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified, aggregate outcome data (summary of OHIP-14 scores, knowledge quiz results, and satisfaction ratings) will be shared. Individual-level raw data will not be shared. Data will be made available in summary tables upon reasonable request for academic purposes, subject to approval by the principal investigator and the Institutional Review Board.